CLINICAL TRIAL: NCT06590584
Title: Validity and Reliability of the 6-minute Pegboard Ring Test in Obese Individuals
Status: Recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_PegboardRingTest
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obese Patients; Obesity; Obese
Keywords: obesity; exercise test; upper extremity; arm exercise endurance
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patients with obesity — Six-Minute Pegboard and Ring Test: It will be used to evaluate upper extremity exercise capacity. There are 20 rings on 4 iron bars on the board used and patients will be asked to attach the rings with both hands, first from top to bottom and then from bottom to top. At the end of the six minutes, the total number of rings attached will be recorded. Heart rate, blood pressure, respiratory rate, dyspnea and fatigue will be evaluated according to the Modified Borg Scale before and after the test.

SUMMARY:
Obesity is a major public health problem that causes numerous diseases and problems that threaten human health. The prevalence of obesity has increased worldwide in the last ~50 years and has reached pandemic levels. Similar results are seen in Turkey, and according to the results of the Turkey Health Survey, 20.2% of people aged 15 and over were obese and 35.6% were pre-obese in 2022. Obesity represents a major health problem as it significantly increases the risk of diseases such as type 2 diabetes mellitus, fatty liver disease, hypertension, myocardial infarction, stroke, dementia, osteoarthritis, obstructive sleep apnea and various cancers, thus contributing to a decrease in both quality of life and life expectancy. Obesity is also associated with unemployment, social disadvantages and reduced socio-economic productivity, thus representing an increasing economic burden.

Obesity is associated with physiological changes at the muscle level, including a decrease in capillary density and blood flow, thus limiting the supply of oxygen and energy resources. Along with the limited blood flow, muscle cells in obese individuals have a decrease in the relative number and size of mitochondria required for energy supply. This leads to a limitation in upper limb activities.

This activity restriction is related to many activities of daily living that involve unsupported upper extremity movements that lead to dyspnea and fatigue in patients with cardiopulmonary disease. Therefore, determining the strength, endurance and exercise capacity of the upper extremities emerges as an important issue in obesity management. One of the tests that serve this purpose is the 6-minute pegboard ring test (6PBRT), which has been found to be valid and reliable in patients with chronic obstructive pulmonary disease and asthma. However, when the literature is examined, it is seen that 6PBRT has not been studied in obese individuals. Therefore, the aim of the study is to investigate the validity and reliability of 6PBRT in obese individuals.

The main question it aims to answer is:

- Is 6PBRT a valid and reliable method to assess upper extremity functional capacity in patients wit obesity?

DETAILED DESCRIPTION:
It was planned as a non-invasive reliability study. The validity and reliability of 6PBRT in obese individuals will be investigated within the scope of the study. In this context, a 1-hour rest break will be given after the first test. Dyspnea and fatigue will be evaluated using the Borg scale and muscle oxygenation, heart rate and blood pressure will be recorded before and after 6PBRT. The second trial of 6PBRT will be performed after the 1-hour rest period. In order to ensure that the patients are stable, the level of dyspnea and fatigue and the initial values of heart rate will be checked before the second trial. All evaluations will be made by the same physiotherapist and an expert physiotherapist will be present during the evaluations.

The smallest sample size of the study was found to be 40 people with a correlation coefficient of 0.95 between the two tests and 90% power at a 95% confidence interval. It is aimed to include 50 people against a 20% drop-out risk.

Shapiro-Wilk test and histogram graphics will be used to check the normality of the data. Demographic and clinical characteristics of the participants will be reported using descriptive statistics. Intraclass correlation coefficient (ICC) with two-way random effects and absolute agreement methods will be used to assess test-retest reliability. The strength of reliability will be interpreted as excellent for ICC value &gt;0.90. Ninety-five percent Confidence Interval (95% CI) will be calculated to investigate measurement variability.

ELIGIBILITY:
Inclusion Criteria:

* BMI value of 30 kg/m2 and above,
* Ability to ambulate,
* Being 18 years of age and above,
* Being a volunteer.

Exclusion Criteria:

* Use of anti-obesity medication,
* Pregnancy,
* Latent autoimmune diabetes,
* Chronic renal failure,
* Active or serious infections,
* Liver failure,
* Recent major cardiovascular events,
* Unstable angina,
* Heart failure (NYHA III-IV)
* Respiratory failure, cardiac arrhythmias, neoplastic diseases, and neurological or musculoskeletal disorders that limit testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese individuals applying to Selçuk University Nutrition and Dietetics Department: Purposive sampling
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Pegboard and Ring Test | 1 hour
  Used to evaluate upper extremity exercise capacity. There are 20 rings on 4 iron bars on the board used, and patients are asked to attach the rings with both hands, first from top to bottom and then from bottom to top. At the end of six minutes, the total number of rings attached is recorded. Before and after the test, heart rate, blood pressure, respiratory rate, dyspnea and fatigue will be evaluated according to the Modified Borg Scale.

SECONDARY OUTCOMES:
Demographic data and personal characteristics | Baseline
  Demographic information such as sociodemographic characteristics and medications used, comorbidities, education level, occupation, smoking and alcohol use, CV and family history of the individuals included in the study will be recorded in a previously prepared form.
Body composition | Baseline
  Body mass and body composition will be measured with the help of Tanita brand device using bioelectrical impedance method. The variables to be evaluated with this device are; body mass index (BMI = body mass: (kg)/height2 (m)2), fat mass expressed as a percentage of body mass (pFM), fat-free mass (FFM) expressed in kilograms and appendicular skeletal muscle mass (ASMM) and skeletal muscle mass (SMM) expressed in kilograms. The measurements will be recorded on the previously prepared form.
Respiratory muscle strength | Baseline
  They are easy to apply and simple measurements. Maximal voluntary inspiratory and expiratory pressures (MIP and MEP) are the most commonly used noninvasive methods for measuring respiratory muscle strength. They are based on the Müller (maximal inspiration) and Valsalva (maximal expiration) principles. MIP and MEP data will be measured and collected with an intraoral pressure measuring device and the data will be recorded on a previously prepared form.
Extremity Muscle Strength | Baseline
  Hand grip, elbow flexion, shoulder flexion and abduction muscle strengths will be measured with a dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulzebos E, Takken T, Reijneveld EA, Mulder MMG, Bongers BC. Reference Values for Respiratory Muscle Strength in Children and Adolescents. Respiration. 2018;95(4):235-243. doi: 10.1159/000485464. Epub 2018 Jan 17. PMID 29342462
- [Background] Zhan S, Cerny FJ, Gibbons WJ, Mador MJ, Wu YW. Development of an unsupported arm exercise test in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2006 May-Jun;26(3):180-7; discussion 188-90. doi: 10.1097/00008483-200605000-00013. PMID 16738459
- [Background] Ozsoy I, Ozcan Kahraman B, Ozsoy G, Ilcin N, Kahraman T, Acar S, Tekin N, Savci S. Determinants of the 6-minute pegboard and ring test as an unsupported upper-extremity exercise capacity measure in older adults with chronic obstructive pulmonary disease. Eur Geriatr Med. 2018 Dec;9(6):863-870. doi: 10.1007/s41999-018-0111-x. Epub 2018 Sep 25. PMID 34674474
- [Background] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557
- [Background] Greco F, Tarsitano MG, Cosco LF, Quinzi F, Folino K, Spadafora M, Afzal M, Segura-Garcia C, Maurotti S, Pujia R, Pujia A, Buono P, Emerenziani GP. The Effects of Online Home-Based Pilates Combined with Diet on Body Composition in Women Affected by Obesity: A Preliminary Study. Nutrients. 2024 Mar 21;16(6):902. doi: 10.3390/nu16060902. PMID 38542813
- [Background] Cavuoto LA, Nussbaum MA. The influences of obesity and age on functional performance during intermittent upper extremity tasks. J Occup Environ Hyg. 2014;11(9):583-90. doi: 10.1080/15459624.2014.887848. PMID 24484265
- [Background] Calik-Kutukcu E, Tekerlek H, Bozdemir-Ozel C, Karaduz BN, Cakmak A, Inal-Ince D, Saglam M, Vardar-Yagli N, Sonbahar-Ulu H, Firat M, Arikan H, Kaya SB, Karakaya G. Validity and reliability of 6-minute pegboard and ring test in patients with asthma. J Asthma. 2022 Jul;59(7):1387-1395. doi: 10.1080/02770903.2021.1930040. Epub 2021 May 31. PMID 33985406
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- See also: Türkiye Health Survey data — https://data.tuik.gov.tr/Bulten/Index?p=Turkiye-Saglik-Arastirmasi-2022-49747